CLINICAL TRIAL: NCT02845986
Title: Safety and Feasibility of Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for Locally Advanced Upper Third Gastric Cancer: A Multicenter Phase II Trial
Brief Title: Study on Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for Advanced Gastric Cancer
Acronym: CLASS-04
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Southwest Hospital, China (Other); Fujian Provincial Hospital (Other); Zhangzhou Municipal Hospital of Fujian Province (Other); Shanghai Zhongshan Hospital (Other); Meizhou People's Hospital (Other); Guangdong Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Second Hospital of Jilin University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Affiliated Hospital of Qinghai University (Other); The First Affiliated Hospital of Xiamen University (Other); RenJi Hospital (Other); West China Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The First Hospital of Putian City, Putian, Fujian (Other Government); Longyan City First Hospital (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University Union Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2016-07-15; First posted 2016-07-27 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopy; Spleen-Preserving; No.10 Lymph Node Dissection
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No.10 lymph node dissections (Experimental): Patients with locally advanced upper third gastric carcinoma will performed laparoscopic spleen-preserving No.10 lymph node dissections.After the surgery the patients will be treated with oxaliplatin or platinum-based chemotherapy.
  Interventions: Procedure: Laparoscopic Spleen-Preserving No.10 Lymph Node Dissections; Drug: oxaliplatin

INTERVENTIONS:
Procedure: Laparoscopic Spleen-Preserving No.10 Lymph Node Dissections — After exclusion of T4b, bulky lymph nodes, or distant metastasis case et al. Laparoscopic spleen-preserving No.10 lymph node dissections will be performed with curative treated intent in patients with locally advanced upper third gastric adenocarcinoma.
Drug: oxaliplatin — oxaliplatin or platinum-based chemotherapy is used when the patients undergo adjuvant chemotherapy after the surgery.
  Other Names: platinum-based chemotherapy

SUMMARY:
The purpose of this study is to explore the safety and feasibility of the Laparoscopic Spleen-Preserving No. 10 Lymph Node Dissection for patients with locally advanced upper third gastric adenocarcinoma（cT2-4a, N-/+, M0）.

DETAILED DESCRIPTION:
Radical resection is still the primary method of treating advanced gastric cancer.According to the Japanese treatment guidelines for gastric cancer, D2 lymphadenectomy, including No. 10 lymph node dissection, should be adopted for upper third gastric carcinoma.The incidence of No. 10 lymph node metastasis is high in advanced proximal gastric cancer, reported to range from 9.8%-20.9%, and the presence of No. 10 lymph node metastasis is closely related to survival. Therefore, in East Asia, D2 lymph node dissection of potentially curable locally advanced upper third gastric cancer including No. 10 lymph node is the standard surgical treatment.

In the early, splenectomy was performed to remove No. 10 lymph node. With the improvement of medical knowledge and surgical technique, spleen-preserving No. 10 lymph node dissection has been recognized by more and more surgeons. However, due to the special and complex anatomy of the spleen, spleen-preserving No. 10 lymph node dissection is difficult, even in open surgery; consequently, the surgery cannot be performed in many centers.

Laparoscopic surgery has distinct minimally invasive advantages, such as small incisions, less blood loss, less postoperative pain, mild postoperative inflammatory reactions, a quick recovery of gastrointestinal function, shorter hospital stays and obvious cosmetic effects. Since Kitano et al. first reported laparoscopic gastrectomy for gastric cancer in 1994, laparoscopic techniques have developed rapidly. The techniques are becoming increasingly mature, making it possible to perform laparoscopic spleen-preserving No. 10 lymph node dissection. Our center first proposed "Huang's three-step maneuver", a new operative method suitable for laparoscopic spleen-preserving No. 10 lymph node dissection. This method simplifies the procedure of laparoscopic spleen-preserving No. 10 lymph node dissection and facilitates its popularization and promotion.

However, it remains a controversial international issue if it is safe and feasible to routinely conduct laparoscopic spleen-preserving No. 10 lymph node dissection for advanced upper third gastric cancer.A number of retrospective studies have successively confirmed the safety, feasibility and oncological efficacy of laparoscopic spleen-preserving No. 10 lymph node dissection.But there is no multicenter prospective studies to identify the results.

Therefore, The study is through a prospective, multicenter, open, single-arm, non-inferiority study,to explore the safety and feasibility of the laparoscopic spleen-preserving No. 10 lymph node dissection for patients with locally advanced upper third gastric adenocarcinoma（cT2-4a, N-/+, M0）.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. Locally advanced tumor in the upper third stomach（cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC(American Joint Committee on Cancer) Cancer Staging Manual Seventh Edition）
4. No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
5. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Written informed consent

Exclusion Criteria:

1. Pregnant and lactating women
2. Suffering from severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous gastric surgery (including ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
5. Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging including enlarged or bulky No.10 lymph node
6. History of other malignant disease within the past 5 years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within the past 6 months
9. History of cerebrovascular accident within the past 6 months
10. History of continuous systematic administration of corticosteroids within 1 month
11. Requirement of simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1<50% of the predicted values
14. Splenectomy must be performed due to the obvious tumor invasion in spleen or spleen blood vessels.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2020-10-12 (Estimated)

PRIMARY OUTCOMES:
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
Numbers of No.10 lymph node dissection | 9 days
  Numbers of dissected No.10 lymph nodes
Rates of positive No.10 lymph node | 9 days
  The Rates of positive No.10 lymph node are defined as the incidence of positive No.10 lymph node (divide number of positive No.10 lymph nodes by number of total No.10 lymph nodes).
3-year overall survival rate | 36 months
3-year disease free survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Rates of splenectomy | 1 days
  The Rates of splenectomy are defined as the incidence of splenectomy within operation.
Intraoperative morbidity rates | 1 days
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
Postoperative pain | 30 days
  Visual analog pain score method is used to evaluate the difference of postoperative pain degree.The score of postoperative pain is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of cholesterol | 3, 6, 9 and 12 months
  The variation of cholesterol in millimole/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of album | 3, 6, 9 and 12 months
  The variation of album in gram/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The results of endoscopy | 3 and 12 months
  The incidence of reflux esophagitis under the endoscopy on postoperative 3 and 12 months are used to access the postoperative quality of life.
The variation of body temperature | 8 days
  The daily highest body temperature in degree centigrade before discharge are recorded to access the inflammatory and immune response.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of prealbumin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of prealbumin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital,China
Locations (20):
- China (20):
  - Beijing Cancer Hospital, Haidian, Beijing Municipality
  - Southwest Hospital, Shapingba, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Longyan First Hospital, Longyan, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Jiangsu province hospital, Nanjing, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Pudong, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Xuhui, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang, Xinjiang

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.

REFERENCES:
- [Result] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2010 (ver. 3). Gastric Cancer. 2011 Jun;14(2):113-23. doi: 10.1007/s10120-011-0042-4. No abstract available. PMID 21573742
- [Result] Monig SP, Collet PH, Baldus SE, Schmackpfeffer K, Schroder W, Thiele J, Dienes HP, Holscher AH. Splenectomy in proximal gastric cancer: frequency of lymph node metastasis to the splenic hilus. J Surg Oncol. 2001 Feb;76(2):89-92. doi: 10.1002/1096-9098(200102)76:23.0.co;2-i. PMID 11223832
- [Result] Chikara K, Hiroshi S, Masato N, Goro M, Yuichi O, Hidetaka O, Hirotoshi A. Association of the number of metastatic perigastric lymph nodes with long-term survival in gastric cancer. Hepatogastroenterology. 2005 Jan-Feb;52(61):277-80. PMID 15783049
- [Result] Bonenkamp JJ, Hermans J, Sasako M, van de Velde CJ, Welvaart K, Songun I, Meyer S, Plukker JT, Van Elk P, Obertop H, Gouma DJ, van Lanschot JJ, Taat CW, de Graaf PW, von Meyenfeldt MF, Tilanus H; Dutch Gastric Cancer Group. Extended lymph-node dissection for gastric cancer. N Engl J Med. 1999 Mar 25;340(12):908-14. doi: 10.1056/NEJM199903253401202. PMID 10089184
- [Result] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Result] Hyung WJ, Lim JS, Song J, Choi SH, Noh SH. Laparoscopic spleen-preserving splenic hilar lymph node dissection during total gastrectomy for gastric cancer. J Am Coll Surg. 2008 Aug;207(2):e6-11. doi: 10.1016/j.jamcollsurg.2008.04.027. No abstract available. PMID 18656040
- [Result] Okabe H, Obama K, Kan T, Tanaka E, Itami A, Sakai Y. Medial approach for laparoscopic total gastrectomy with splenic lymph node dissection. J Am Coll Surg. 2010 Jul;211(1):e1-6. doi: 10.1016/j.jamcollsurg.2010.04.006. No abstract available. PMID 20610241
- [Result] Hur H, Jeon HM, Kim W. Laparoscopic pancreas- and spleen-preserving D2 lymph node dissection in advanced (cT2) upper-third gastric cancer. J Surg Oncol. 2008 Feb 1;97(2):169-72. doi: 10.1002/jso.20927. PMID 18095269
- [Result] Schwarz RE. Spleen-preserving splenic hilar lymphadenectomy at the time of gastrectomy for cancer: technical feasibility and early results. J Surg Oncol. 2002 Jan;79(1):73-6. doi: 10.1002/jso.10036. No abstract available. PMID 11754382
- [Result] Tanimura S, Higashino M, Fukunaga Y, Kishida S, Ogata A, Fujiwara Y, Osugi H. Laparoscopic gastrectomy with regional lymph node dissection for upper gastric cancer. Br J Surg. 2007 Feb;94(2):204-7. doi: 10.1002/bjs.5542. PMID 17058319
- [Result] Huang CM, Chen QY, Lin JX, Zheng CH, Li P, Xie JW. Huang's three-step maneuver for laparoscopic spleen-preserving No. 10 lymph node dissection for advanced proximal gastric cancer. Chin J Cancer Res. 2014 Apr;26(2):208-10. doi: 10.3978/j.issn.1000-9604.2014.04.05. PMID 24826062
- [Result] Jung MR, Park YK, Seon JW, Kim KY, Cheong O, Ryu SY. Definition and classification of complications of gastrectomy for gastric cancer based on the accordion severity grading system. World J Surg. 2012 Oct;36(10):2400-11. doi: 10.1007/s00268-012-1693-y. PMID 22752074
- [Result] Orsenigo E, Bissolati M, Socci C, Chiari D, Muffatti F, Nifosi J, Staudacher C. Duodenal stump fistula after gastric surgery for malignancies: a retrospective analysis of risk factors in a single centre experience. Gastric Cancer. 2014 Oct;17(4):733-44. doi: 10.1007/s10120-013-0327-x. Epub 2014 Jan 8. PMID 24399492
- [Result] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Result] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Result] Asgeirsson T, El-Badawi KI, Mahmood A, Barletta J, Luchtefeld M, Senagore AJ. Postoperative ileus: it costs more than you expect. J Am Coll Surg. 2010 Feb;210(2):228-31. doi: 10.1016/j.jamcollsurg.2009.09.028. Epub 2009 Nov 18. PMID 20113944
- [Result] Arozullah AM, Khuri SF, Henderson WG, Daley J; Participants in the National Veterans Affairs Surgical Quality Improvement Program. Development and validation of a multifactorial risk index for predicting postoperative pneumonia after major noncardiac surgery. Ann Intern Med. 2001 Nov 20;135(10):847-57. doi: 10.7326/0003-4819-135-10-200111200-00005. PMID 11712875
- [Result] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Infect Control Hosp Epidemiol. 1992 Oct;13(10):606-8. No abstract available. PMID 1334988
- [Result] Dong K, Yu XJ, Li B, Wen EG, Xiong W, Guan QL. Advances in mechanisms of postsurgical gastroparesis syndrome and its diagnosis and treatment. Chin J Dig Dis. 2006;7(2):76-82. doi: 10.1111/j.1443-9573.2006.00255.x. PMID 16643334
- [Result] Kaas R, Rustman LD, Zoetmulder FA. Chylous ascites after oncological abdominal surgery: incidence and treatment. Eur J Surg Oncol. 2001 Mar;27(2):187-9. doi: 10.1053/ejso.2000.1088. PMID 11289756
- [Result] Assumpcao L, Cameron JL, Wolfgang CL, Edil B, Choti MA, Herman JM, Geschwind JF, Hong K, Georgiades C, Schulick RD, Pawlik TM. Incidence and management of chyle leaks following pancreatic resection: a high volume single-center institutional experience. J Gastrointest Surg. 2008 Nov;12(11):1915-23. doi: 10.1007/s11605-008-0619-3. Epub 2008 Aug 7. PMID 18685899
- [Result] Greenblatt DY, Kelly KJ, Rajamanickam V, Wan Y, Hanson T, Rettammel R, Winslow ER, Cho CS, Weber SM. Preoperative factors predict perioperative morbidity and mortality after pancreaticoduodenectomy. Ann Surg Oncol. 2011 Aug;18(8):2126-35. doi: 10.1245/s10434-011-1594-6. Epub 2011 Feb 20. PMID 21336514
- [Derived] Xu BB, Zheng HL, Chen CS, Xu LL, Xue Z, Wei LH, Zheng HH, Shen LL, Zheng CH, Li P, Xie JW, Lin JX, Zheng YH, Huang CM. Development and validation of a preoperative radiomics-based nomogram to identify patients who can benefit from splenic hilar lymphadenectomy: a pooled analysis of three prospective trials. Int J Surg. 2024 Jul 1;110(7):4053-4061. doi: 10.1097/JS9.0000000000001337. PMID 38980664